CLINICAL TRIAL: NCT00197249
Title: A Phase III, Open, Randomized, Multicentric Study to Compare the Reactogenicity and Immunogenicity of GSK Biologicals' Combined Vi Polysaccharide Typhoid Vaccine and Inactivated Hepatitis A Vaccine, to That Elicited by GSK Biologicals' Hepatitis A Vaccine, Administered Singly or Concomitantly With GSK Biologicals' Vi Polysaccharide Vaccine
Brief Title: Comparative Study in Healthy Adults Aged 18-50 Yrs Administered With Hepatyrix or Havrix+Typherix or Tiphim Vi, to Compare Reactogenicity & Immunogenicity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 270362/006; 270362/007 (Ext. Mth12) (Other: GSK); 270362/008 (Ext. Mth24) (Other: GSK); 270362/009 (Ext. Mth36) (Other: GSK)
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis A
Keywords: Hepatitis A & B; Typhoid
MeSH Terms: conditions — Hepatitis A; Typhoid Fever

INTERVENTIONS:
Biological: Combined Vi polysaccharide typhoid vaccine and hepatitis A vaccine- Hepatyrix

SUMMARY:
To evaluate the immunogenicity, reactogenicity and safety of Hepatyrix when compared to the concomitant administration of Typherix and Havrix, and when compared to the administration of monovalent vaccines, Havrix or Typhim Vi. Furthermore, the study will evaluate the persistence of anti-Vi and anti-HAV antibodies up to 36 months after administration of the first dose of the study vaccine.

DETAILED DESCRIPTION:
Compare the reactogenicity & immunogenicity of GSK Biologicals' combined Vi polysaccharide typhoid vaccine & inactivated hepatitis A vaccine, Hepatyrix, to that elicited by GSK Biologicals' hepatitis A vaccine, Havrix administered singly or concomitantly with GSK Biologicals' Vi polysaccharide vaccine, Typherix, & to that elicited by Aventis Pasteur's monovalent Vi polysaccharide vaccine, Typhim Vi, administered intramuscularly to healthy subjects aged 18-65 yrs.

ELIGIBILITY:
Inclusion criteria

* Written informed consent will be obtained from the subject prior to entry into the study.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Seronegative for anti-HAV antibodies.
* If the subject is female, she must be of non-childbearing potential, i.e., either surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (e.g., intrauterine contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream or foam; Norplant® or DepoProvera®) for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.
* Subjects having received the study vaccines 36 months earlier.

Exclusion criteria

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. (For corticosteroids, this will mean prednisone, or equivalent, >or = 0.5 mg/kg/day. Inhaled and topical steroids are allowed.).
* Planned administration/Administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s).
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* History of chronic alcohol consumption and/or intravenous drug abuse.
* Previous vaccination against hepatitis A.
* Previous vaccination against typhoid fever.
* History of hepatitis A.
* Previous diagnosis, confirmed by a physician, of Salmonella typhi infection.
* History of non-response to hepatitis A and or typhoid vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e., axillary temperature < 99.5 °F (37.5 °C)
* Female planning to become pregnant during the primary study period (up Month 7).
* Pregnant or lactating female.
* Planned travel to areas of high endemicity for hepatitis A and/ or typhoid fever during the primary study period (up Month 7).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1034 (Actual)
Dates: Start 2002-05; Primary Completion 2003-06 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Anti-Vi seropositivity rates (i.e., percentage of subjects with anti-Vi antibody titres > or = 150 EL.U/ml) at Month 1 after administration of study vaccine (Comparison of Hepatyrix versus concomitant Havrix+Typherix and Hepatyrix versus Typhim Vi).
Anti-HAV seropositivity rates (i.e., percentage of subjects with anti-HAV antibody titres >or = 15 mIU/ml) at Month 1 after administration of study vaccine, (Comparison of Hepatyrix versus concomitant Havrix+Typherix and Hepatyrix versus Havrix).

SECONDARY OUTCOMES:
Anti-Vi seropositivity rates at Day 14, Month 6 and Month 7 and GMTs at Day 14, Month 1, Month 6 and Month 7 after administration of study vaccine.
Anti-HAV seropositivity rates at Day 14, Month 6 and Month 7 and GMTs at Day 14, Month 1, Month 6 and Month 7 after administration of study vaccine.
Anti-Vi and anti-HAV seropositivity rates and GMTs at Months 12, 24, 36 after administration of study vaccine.
Occurrence and intensity of solicited local symptoms after vaccination (Day 0 to 4).
Occurrence, intensity and relationship of solicited general symptoms after vaccination (Day 0 to 4).
Occurrence, intensity and relationship to vaccination of unsolicited signs and symptoms after vaccination (Day 0 to 30).
Occurrence, intensity and relationship to vaccination of serious adverse events (SAEs) during the study period and during the follow-up period up to Months 12, 24 and 36 after administration of study vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 270362/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 270362/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 270362/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 270362/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 270362/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register